CLINICAL TRIAL: NCT04072133
Title: Effects of Meditative Movement on Body Composition in Midlife Women
Brief Title: The Move Well Study
Acronym: MW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005974
Record Dates: First submitted 2019-08-13; First posted 2019-08-28 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Effects of Meditative Movement on Body Composition
Keywords: Midlife Women; Body Composition; Meditative Movement; Emotional Eating; Sleep Quality; Body Fat Percentage; Tai Chi Easy
MeSH Terms: conditions — Emotional Eating; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Clinical trial with single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meditative Movement Intervention (Experimental): Participants will complete the following components of baseline (T1) data collection: demographics, biometric measurements, a heart rate variability assessment, and questionnaires. Participants will be asked to provide six saliva samples via passive drool to measure cortisol levels. Participants will be assigned into hour-long meditative movement (MM) classes for eight weeks total. Participants will be asked to practice their MM skills at home for at least 30 minutes most days per week. The study will distribute hard-copy movement manuals and DVD instruction videos for guidance. Participants will be asked to provide a log of all dates and lengths of their at-home practice. After the eighth class, participants will return for post-intervention (T2) data collection, consisting of biometric measurements, a heart rate variability assessment, and questionnaires. Participants will provide six more saliva samples via passive drool method.
  Interventions: Behavioral: Meditative Movement

INTERVENTIONS:
Behavioral: Meditative Movement — Intervention will be taught by a certified Tai Chi Easy (TCE) group practice leader. The TCE movements will be repeated in differing sequences and time-frames during the course of the study. The variety and combination of the exercises will begin easy and progress to more advanced movements and/or intensities as the study progresses and participants become more experienced and comfortable with the routine. Participants spend one hour in class each week for a total of eight weeks.
  Other Names: Tai Chi Easy (TCE)

SUMMARY:
This study will explore the effects of meditative movement on body composition in a group of 60 midlife women. Women will participate in 30-minute meditative movement (MM) classes for an eight-week period. Participants will be encouraged to practice MM at home for at least 30 minutes most days per week. Participants will be asked to complete a log of their time spent doing meditative movement outside of classes.

DETAILED DESCRIPTION:
A growing body of published evidence indicates that meditative movement (MM) practices may be helpful for body composition improvement. Less strenuous forms of exercise that include a focus on the breath and meditative state (i.e., "meditative movement" such as Yoga, Qigong, or Tai Chi) may be easier to adopt for unfit, sedentary, overweight or obese women, which characterizes a large percentage of the general population. Despite this preliminary evidence, no studies have proposed a model for how or why weight loss might occur in MM interventions where the goals are not designated as weight loss, nutritional counseling is not included, and energy expenditure is not at the level assumed to be required to achieve weight loss. The proposed intervention is designed to refine and gather preliminary evidence for a novel "mindful-body-wisdom" model of intervening on improving body composition and to examine the contribution of model factors (psychological and behavioral) of how such a non-diet/non-vigorous exercise intervention might work, in 60 midlife women.

TCE is a simple TC/QG form that was developed by Dr. Roger Jahnke and developed into a standardized research intervention protocol by a team of researchers. It has been used in several prior projects and one recently completed NIH/NCCAM-funded randomized controlled trial (RCT) with breast cancer survivors showing reduction in fatigue and depression, and improved sleep and physical function.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 45-75 years of age
* Ability to participate in low intensity activity

Exclusion Criteria:

* Women who are unable to stand for 10-minute segments (e.g., wheelchair or walker bound and too weak)
* Women who are unable to walk

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be female
Enrollment: 52 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Body Fat Percentage | 8 weeks
  Body fat percentage will be measured using Bioelectric Impedance Analysis (BIA) via the Tanita monitor. Score range= 0% to 100%. A higher score indicates a higher body fat percentage.
Emotional Eating | 8 weeks
  Emotional eating will be measured using the Three Factor Eating Questionnaire (TFEQ) (21 items, 4-point Likert scale with response options 1 through 4 for items 1 through 17, response options 1 through 8 for item 18). Score range= 18 to 76. Emotional eating sub-score is calculated by combining six items of the TFEQ. A higher score indicates greater emotional eating.
Sleep Quality | 8 weeks
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI) (10 items, 4-point Likert scale; 0= positive extreme of scale, 3= negative extreme of scale). Score range= 0 to 21. A higher score indicates worse sleep quality.

SECONDARY OUTCOMES:
Perceived Stress Scale-10 | 8 weeks
  self-report measure of perceived stress, 10-items, Likert scale
Self-Compassion Scale (SCS) | 8 weeks
  self-report measure of self-compassion as measured (26 items) by self-kindness, common humanity, non-judgment
Body Awareness Questionnaire (BAQ) | 8 weeks
  self-report measure of experienced body awareness/iteroception, 18-items, Likert-scale
Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) | 8 weeks
  self-report measure of mindfulness, Likert-scale, 9-items

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University Downtown Campus, Phoenix, Arizona, United States